CLINICAL TRIAL: NCT03644160
Title: A Physiotherapist Led Intervention to Promote Physical Activity in Rheumatoid Arthritis - a Pilot Study
Acronym: PIPPRA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Limerick (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PIPPRA-1
Record Dates: First submitted 2018-05-01; First posted 2018-08-23 (Actual); Last update posted 2022-06-13 (Actual); Status verified 2022-06

CONDITIONS: Rheumatoid Arthritis
Keywords: Physical activity; Behaviour Change; Physiotherapy
MeSH Terms: conditions — Arthritis, Rheumatoid; Motor Activity | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Single-centre randomised pilot study
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Physical activity and behaviour change The intervention group (group A) will receive an 8 week individualised, tailored behaviour change intervention to promote PA and an information booklet about physical activity with a physiotherapist who has training in behaviour change techniques and motivational interviewing. Using a range of behaviour change and self-regulation techniques (eg goal-setting, self-monitoring), participants will be guided towards physical activity maintenance at the end of the 8 weeks. In addition, participants will be signposted to physical activity classes, facilities and resources in the local community. This group will continue with their routine care for their condition throughout the study period.
  Interventions: Behavioral: Physical activity and behaviour change
- Control Group (No Intervention): The control group (Group B) will receive the same information booklet about physical activity only. This group will continue with their routine care for their condition throughout the study period.

INTERVENTIONS:
Behavioral: Physical activity and behaviour change — The intervention group (group A) will receive an 8 week individualised, tailored behaviour change intervention to promote PA and an information booklet about physical activity to include an initial 1:1 session with a physiotherapist with training in behaviour change techniques and motivational interviewing. Using a range of behaviour change and self-regulation techniques (eg goal-setting, self-monitoring), participants will be guided towards physical activity maintenance at the end of the 8 weeks. In addition, participants will be signposted to physical activity classes, facilities and resources in the local community. This group will continue with their routine care for their condition throughout the study period.
  Arms: Intervention Group

SUMMARY:
Rheumatoid arthritis (RA), a chronic, inflammatory condition with increased mortality from cardiovascular disease, is associated with high health care related costs and decreased productivity. Currently, nonpharmacological management guidelines recommend increasing low levels of physical activity in this group to improve health including cardiovascular health, yet research has shown that people who have RA have reduced levels of PA. Interventions targeting PA behaviour in this population have had limited effect to date due to lack of patient involvement in designing the intervention, poor measurement of PA, lack of behaviour change theory underpinning the intervention and have tended to include people who already have some level of PA. Work to underpin a robust intervention to improve PA in this group has been undertaken by members of this study group including validation of an objective measure PA in RA and interviews with people who have RA and rheumatology health professionals to aid in designing an intervention to promote PA.

The aim of this pilot randomised controlled trial (RCT) is to examine the feasibility of a physiotherapist led, behaviour change theory informed, PA intervention to promote PA in people who have RA who have low levels of current PA. This pilot study will determine the rate of recruitment to the study and also determine the acceptability of the intervention to the participants as well as test the feasibility of the secondary disease/PA focused outcome measures.

Participants will be recruited from rheumatology clinics in a large teaching hospital. Participants meeting inclusion criteria will be randomised into an eight week PA intervention (four sessions delivered over an eight week period by a trained physiotherapist) or a control group (PA information leaflet). This pilot randomised study will provide valuable information for the scaling up of a primary care based intervention for this important patient group and in doing so provide an achievable, pragmatic intervention for busy clinicians, who need feasible interventions to appropriately manage complex chronic conditions like RA in a busy primary care setting.

DETAILED DESCRIPTION:
Rheumatoid Arthritis (RA) affects approximately 0.5% of the adult population worldwide. In Ireland c46,000 people have RA, with c2,000 new cases diagnosed annually. Cardiovascular disease (CVD) , infections and lymphoma occur more frequently in this population with increased mortality rates present1. Physical activity (PA) is very important in the management of RA and is an essential in reducing the risk of CVD, improving disease symptoms and quality of life. However, people who have RA tend to have low PA levels, thus improving PA levels is important. Previous interventions which have targeted PA in people who have RA have had limited success in increasing and maintaining PA behaviour change (BC) in the longer term. Reasons for this limited success include short intervention time, inadequate involvement of participants in designing the study, lack of objective measurement of PA and lack of a BC theoretical underpinning. Thus, better intervention design through the incorporation of appropriate BC theory is necessary. Adopting the Behaviour Change Wheel (BCW), facilitates the identification of factors which should be targeted in a BC intervention to promote PA. In order to design a robust intervention to address the issues above, the applicants undertook extensive systematic literature reviewing, objective PA measurement validation and qualitative interviews with people with RA and with rheumatology health professionals, guided by the Medical Research council framework for complex interventions. A pilot intervention is now proposed building on that work to determine the feasibility of a physiotherapist led BC intervention to promote PA in people with RA who have low levels of PA.

The aim of this pilot study is to determine the feasibility and acceptability of a physiotherapist led BC intervention to promote PA in people with RA who are insufficiently physically active compared to a control group who receive a leaflet on PA.

Ethical Approval: approval will be sought in advance of the study start date from Health Service Executive Research ethics committee University Hospitals Limerick.

Trial design: single-centre randomised pilot study, incorporating qualitative interviews to examine acceptability, comparing the intervention with a control.

Methods: Participants, interventions, and outcomes Study setting - Academic teaching hospitals group in Mid-West of Ireland

Interventions The intervention group (group A) will receive an 8 week individualised, tailored behaviour change intervention to promote PA and an information booklet about PA with a physiotherapist with training in behaviour change techniques and motivational interviewing. Using a range of behaviour change and self-regulation techniques (eg goal-setting, self-monitoring), participants will be guided towards PA maintenance at the end of the 8 weeks. In addition, participants will be signposted to PA classes, facilities and resources in the local community.

The control group (Group B) will receive the same information booklet about PA only. Both groups will continue with their routine care for their condition throughout the study period.

Primary outcome measures will be:

1. Recruitment rate - the rate of participants recruited to the study versus total potential participants
2. Retention rate - the number of participants who complete baseline measures and at week 8

Sample Size A target of 40 participants, with 20 participants in both the control and intervention groups. This sample size is expected to provide sufficient data to meet the primary outcomes. A definitive sample size of a large-scale RCT will be determined from the results of this trial.

Data analysis Descriptive statistics will be used to determine the recruitment and retentions rates and to measure change in outcome measures from baseline to T1 and T2. Thematic analysis will be used to analyse the transcribed interviews

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Rheumatoid arthritis
* Age over 18 years
* Classified using Godin-Shephard Leisure-Time Physical Activity Questionnaire as insufficiently active

Exclusion Criteria:

* Aged less than 18 years
* People who require a mobility aid to mobilise in their activities of daily living (ADLs)
* Pregnancy
* Meeting aerobic physical activity recommendations already

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2021-11-01 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Recruitment rate | Baseline
  The rate of participants recruited to the study versus total potential participants
Retention rate | At week 12
  The number of participants who complete baseline measures at week 12

SECONDARY OUTCOMES:
Physical activity - objective | Baseline, 8 and 24-week follow-up
  Physical activity profile measured using accelerometry (ActivPal)
Physical activity - self-report | Baseline, 8 and 24-week follow-up
  Self report physical activity (Yale Physical Activity Survey)
Behaviour Change | Baseline, 8 and 24-week follow-up
  Theory of planned behaviour questionnaire (TPBQ)
Quality of Life in Rheumatoid Arthritis | Baseline, 8 and 24-week follow-up
  Quality of Life in Rheumatoid Arthritis (RAQoL) will be used to examine self-reported quality of life in rheumatoid arthritis
Pain over past 7 days | Baseline, 8 and 24-week follow-up
  Visual analogue scale (VAS) will measure self-reported pain levels. 100 mm VAS from 0 (no pain) to 100 (most possible pain).
Fatigue | Baseline, 8 and 24-week follow-up
  Bristol RA Fatigue Multi-dimensional Questionnaire (BRAF-MDQ)
Function | Baseline, 8 and 24-week follow-up
  Health assessment questionnaire (HAQ)
Sleep | Baseline, 8 and 24-week follow-up
  Pittsburgh Sleep Quality Index
Disease activity profile | Baseline, 8 and 24-week follow-up
  The Disease Activity Score 28 (DAS28) combines single measures into an overall, continuous measure of rheumatoid arthritis (RA) disease activity. The DAS28 includes a 28 tender joint count, a 28 swollen joint count, erythrocyte sedimentation rate, and a general health assessment on a visual analog scale.

CONTACTS AND LOCATIONS:
Overall Officials: Norelee Kennedy, PhD, Principal Investigator — University of Limerick
Locations (1):
- University of Limerick/University Hospitals Limerick, Limerick, Ireland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Carmona L, Cross M, Williams B, Lassere M, March L. Rheumatoid arthritis. Best Pract Res Clin Rheumatol. 2010 Dec;24(6):733-45. doi: 10.1016/j.berh.2010.10.001. PMID 21665122
- [Background] Power D, Codd M, Ivers L, Sant S, Barry M. Prevalence of rheumatoid arthritis in Dublin, Ireland: a population based survey. Ir J Med Sci. 1999 Jul-Sep;168(3):197-200. doi: 10.1007/BF02945853. PMID 10540788
- [Background] Peters MJ, Symmons DP, McCarey D, Dijkmans BA, Nicola P, Kvien TK, McInnes IB, Haentzschel H, Gonzalez-Gay MA, Provan S, Semb A, Sidiropoulos P, Kitas G, Smulders YM, Soubrier M, Szekanecz Z, Sattar N, Nurmohamed MT. EULAR evidence-based recommendations for cardiovascular risk management in patients with rheumatoid arthritis and other forms of inflammatory arthritis. Ann Rheum Dis. 2010 Feb;69(2):325-31. doi: 10.1136/ard.2009.113696. Epub 2009 Sep 22. PMID 19773290
- [Background] Cooney JK, Law RJ, Matschke V, Lemmey AB, Moore JP, Ahmad Y, Jones JG, Maddison P, Thom JM. Benefits of exercise in rheumatoid arthritis. J Aging Res. 2011 Feb 13;2011:681640. doi: 10.4061/2011/681640. PMID 21403833
- [Background] Swardh E, Brodin N. Effects of aerobic and muscle strengthening exercise in adults with rheumatoid arthritis: a narrative review summarising a chapter in Physical activity in the prevention and treatment of disease (FYSS 2016). Br J Sports Med. 2016 Mar;50(6):362-7. doi: 10.1136/bjsports-2015-095793. Epub 2016 Feb 3. PMID 26843536
- [Background] Sokka T, Hakkinen A, Kautiainen H, Maillefert JF, Toloza S, Mork Hansen T, Calvo-Alen J, Oding R, Liveborn M, Huisman M, Alten R, Pohl C, Cutolo M, Immonen K, Woolf A, Murphy E, Sheehy C, Quirke E, Celik S, Yazici Y, Tlustochowicz W, Kapolka D, Skakic V, Rojkovich B, Muller R, Stropuviene S, Andersone D, Drosos AA, Lazovskis J, Pincus T; QUEST-RA Group. Physical inactivity in patients with rheumatoid arthritis: data from twenty-one countries in a cross-sectional, international study. Arthritis Rheum. 2008 Jan 15;59(1):42-50. doi: 10.1002/art.23255. PMID 18163412
- [Background] Tierney M, Fraser A, Kennedy N. Physical activity in rheumatoid arthritis: a systematic review. J Phys Act Health. 2012 Sep;9(7):1036-48. doi: 10.1123/jpah.9.7.1036. PMID 22971883
- [Background] Brodin N, Hurkmans E, DiMatteo L, Nava T, Vliet Vlieland T, Opava CH. Promotion of health-enhancing physical activity in rheumatoid arthritis: a comparative study on healthcare providers in Italy, The Netherlands and Sweden. Rheumatol Int. 2015 Oct;35(10):1665-73. doi: 10.1007/s00296-015-3267-4. Epub 2015 Apr 14. PMID 25869348
- [Background] Knittle K, De Gucht V, Hurkmans E, Peeters A, Ronday K, Maes S, Vlieland TV. Targeting motivation and self-regulation to increase physical activity among patients with rheumatoid arthritis: a randomised controlled trial. Clin Rheumatol. 2015 Feb;34(2):231-8. doi: 10.1007/s10067-013-2425-x. Epub 2013 Nov 9. PMID 24213780
- [Background] Larkin L, Gallagher S, Cramp F, Brand C, Fraser A, Kennedy N. Behaviour change interventions to promote physical activity in rheumatoid arthritis: a systematic review. Rheumatol Int. 2015 Oct;35(10):1631-40. doi: 10.1007/s00296-015-3292-3. Epub 2015 May 21. PMID 25994094
- [Background] Larkin L, Nordgren B, Purtill H, Brand C, Fraser A, Kennedy N. Criterion Validity of the activPAL Activity Monitor for Sedentary and Physical Activity Patterns in People Who Have Rheumatoid Arthritis. Phys Ther. 2016 Jul;96(7):1093-101. doi: 10.2522/ptj.20150281. Epub 2015 Dec 4. PMID 26637646
- [Background] Larkin L, Gallagher S, Fraser A, Kennedy N. If a joint is hot it's not the time: health professionals' views on developing an intervention to promote physical activity in rheumatoid arthritis. Disabil Rehabil. 2017 Jun;39(11):1106-1113. doi: 10.1080/09638288.2016.1180548. Epub 2016 Jun 8. PMID 27278440
- [Background] Larkin L, Kennedy N, Fraser A, Gallagher S. 'It might hurt, but still it's good': People with rheumatoid arthritis beliefs and expectations about physical activity interventions. J Health Psychol. 2017 Nov;22(13):1678-1690. doi: 10.1177/1359105316633286. Epub 2016 Mar 8. PMID 26962132
- [Background] Michie S, van Stralen MM, West R. The behaviour change wheel: a new method for characterising and designing behaviour change interventions. Implement Sci. 2011 Apr 23;6:42. doi: 10.1186/1748-5908-6-42. PMID 21513547
- [Derived] Larkin L, McKenna S, Pyne T, Comerford P, Moses A, Folan A, Gallagher S, Glynn L, Fraser A, Esbensen BA, Kennedy N. Promoting physical activity in rheumatoid arthritis through a physiotherapist led behaviour change-based intervention (PIPPRA): a feasibility randomised trial. Rheumatol Int. 2024 May;44(5):779-793. doi: 10.1007/s00296-024-05544-1. Epub 2024 Mar 4. PMID 38438576